CLINICAL TRIAL: NCT06764576
Title: Epidemiological, Demographic and Clinical Aspects of Patients With Tuberculosis, Mycobacteriosis or Infection Latent Tuberculosis
Brief Title: Patients With Tuberculosis, Mycobacteriosis or Latent Tuberculosis
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Micro-TB
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Mycobacterial Infection; Tuberculosis (TB)
Keywords: infection; mycobacterial; tuberculosis; diagnosis; latent tuberculosis infection; mycobacterial non-tubercular; microbiological tests
MeSH Terms: conditions — Mycobacterium Infections; Tuberculosis; Infections; Disease; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood, sputum or broncholavage samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tuberculosis or mycobacteriosis Microbiologically confirmed cases: Retrospective phase from 1 January 2012 to 31 May 2021
- Latent tuberculosis infection cases: Retrospective phase, patients followed by infectious diseases clinics from 2017 to May 2021
- Patients with suspected tuberculosis, non-tubercular mycobacteriosis or tubercular infection: Prospective phase from 1 June 2021 to 31 December 2026

SUMMARY:
In the last 30 years, tuberculosis (TB) has re-emerged in industrialised countries as a public health, with a decrease in incidence among the resident population and an increase in the burden of immigrants. Therefore, it becomes a priority to implement an effective TB control that relies on both rapid and reliable identification of active infections, with a adequate treatment and surveillance of resistance, but also on the identification of latent tuberculosis infections (ITBL) in populations at higher risk of progression to the active disease, representing a source of infection for the community.

DETAILED DESCRIPTION:
The study is non-pharmacological and monocentric. Data from patients with clinical/radiological suspicion of mycobacteriosis or tuberculosis will be considered for which they have been received at the OU of Microbiology of the Polyclinic S.Orsola-Malpighi biological samples for mycobacteria research and/or blood samples for immunological investigations for latent tubercular infection in the period January 2012-May 2021 (retrospective part of the study); Data from patients suspected of mycobacteriosis, TB or ITBL from June 2021 to December 2026 (prospective part of the study, duration: 6 years, possibly renewable) will also be considered. The objectives of the study are: 1) Analysis of epidemiological, demographic and clinical aspects of patients with TB, mycobacteriosis non-tubercular or ITBL in the period January 2012-December 2026. 2) Assessment of diagnostic accuracy of the most frequently used methods for Microbiological diagnosis of tuberculosis (TB) or non-tubercular mycobacteriosis and immunological methods for the diagnosis of latent tubercular infection (ITBL). 3) Analysis of the microbiological characteristics (phenotypic and molecular) of MTB and NTM strains. 4) Evaluation of the clinical outcome of patients with ITBL/TB/NTM in treatment and follow-up in the post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 years or more,
* clinical/radiological suspicion of TB or non-tubercular mycobacteriosis or ITBL for which sent to the Microbiology laboratory at least one biological sample for the mycobacteria and/or a blood sample for the IGRA test;
* Obtaining informed consent.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the retrospective phase: TB or mycobacteriosis cases confirmed and ITBL cases followed by Infectious Disease Unit.
  For the prospective phase: TB, non-tubercular mycobacteriosis or ITBL patients with suspicion.
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Estimated)
Dates: Start 2021-12-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of epidemiological, demographic and clinical aspects of patients with tuberculosis, mycobacteriosis non-tubercular or latent tubercular infection | from 2021 to 2026
  Patients' data with biological samples for mycobacteria research and/or blood samples for immunological investigations for latent tubercular infection and clinical/radiological suspicion of mycobacteriosis or tuberculosis had been colleted from January 2012 to May 2021 (retrospective phase of the study) and from June 2021 to December 2026 (prospective phase of the study). The criteria for diagnosis of TB confirmed microbiologically are: Clinical+Imaging suggestive of tuberculosis disease;microbiological isolation of MTB and/ or molecular test for MTB (Xpert) positive;decision of the clinician to start anti-tuberculosis treatment. The criteria for diagnosing non-tubercular mycobacteriosis are: Clinical+Imaging suggestive of mycobacteriosis;isolation of NTM from at least two sputum samples or one bronchocolagement sample. The criteria for diagnosing ITBL are: positive IGRA and/or positive TST test;absence of clinical/radiological signs of tubercular disease.

SECONDARY OUTCOMES:
Assessment of the diagnostic accuracy of the most frequently used methods for microbiological diagnosis of tuberculosis (TB) or non-tubercular mycobacteriosis and Immunological methods for the diagnosis of latent tubercular infection (ITBL). | from 2021 to 2026
  Patients' data with biological samples for mycobacteria research and/or blood samples for immunological investigations for latent tubercular infection and clinical/radiological suspicion of mycobacteriosis or tuberculosis had been colleted from January 2012 to May 2021 (retrospective phase of the study) and from June 2021 to December 2026 (prospective phase of the study). The criteria for diagnosis of TB confirmed microbiologically are: Clinical+Imaging suggestive of tuberculosis disease;microbiological isolation of MTB and/ or molecular test for MTB (Xpert) positive;decision of the clinician to start anti-tuberculosis treatment. The criteria for diagnosing non-tubercular mycobacteriosis are: Clinical+Imaging suggestive of mycobacteriosis;isolation of NTM from at least two sputum samples or one bronchocolagement sample. The criteria for diagnosing ITBL are: positive IGRA and/or positive TST test;absence of clinical/radiological signs of tubercular disease.

OTHER OUTCOMES:
Analysis of the microbiological characteristics (phenotypic and molecular) of MTB and NTM. | from 2021 to 2026
  Patients' data with biological samples for mycobacteria research and/or blood samples for immunological investigations for latent tubercular infection and clinical/radiological suspicion of mycobacteriosis or tuberculosis had been colleted from January 2012 to May 2021 (retrospective phase of the study) and from June 2021 to December 2026 (prospective phase of the study). The criteria for diagnosis of TB confirmed microbiologically are: Clinical+Imaging suggestive of tuberculosis disease;microbiological isolation of MTB and/ or molecular test for MTB (Xpert) positive;decision of the clinician to start anti-tuberculosis treatment. The criteria for diagnosing non-tubercular mycobacteriosis are: Clinical+Imaging suggestive of mycobacteriosis;isolation of NTM from at least two sputum samples or one bronchocolagement sample. The criteria for diagnosing ITBL are: positive IGRA and/or positive TST test;absence of clinical/radiological signs of tubercular disease.
Evaluation of the clinical outcome of patients with ITBL/TB/NTM in treatment and follow-up in post-processing period. | from 2021 to 2026
  Patients' data with biological samples for mycobacteria research and/or blood samples for immunological investigations for latent tubercular infection and clinical/radiological suspicion of mycobacteriosis or tuberculosis had been colleted from January 2012 to May 2021 (retrospective phase of the study) and from June 2021 to December 2026 (prospective phase of the study). The criteria for diagnosis of TB confirmed microbiologically are: Clinical+Imaging suggestive of tuberculosis disease;microbiological isolation of MTB and/ or molecular test for MTB (Xpert) positive;decision of the clinician to start anti-tuberculosis treatment. The criteria for diagnosing non-tubercular mycobacteriosis are: Clinical+Imaging suggestive of mycobacteriosis;isolation of NTM from at least two sputum samples or one bronchocolagement sample. The criteria for diagnosing ITBL are: positive IGRA and/or positive TST test;absence of clinical/radiological signs of tubercular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Dal Monte, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haworth CS, Banks J, Capstick T, Fisher AJ, Gorsuch T, Laurenson IF, Leitch A, Loebinger MR, Milburn HJ, Nightingale M, Ormerod P, Shingadia D, Smith D, Whitehead N, Wilson R, Floto RA. British Thoracic Society guidelines for the management of non-tuberculous mycobacterial pulmonary disease (NTM-PD). Thorax. 2017 Nov;72(Suppl 2):ii1-ii64. doi: 10.1136/thoraxjnl-2017-210927. No abstract available. PMID 29054853
- [Background] Nahid P, Dorman SE, Alipanah N, Barry PM, Brozek JL, Cattamanchi A, Chaisson LH, Chaisson RE, Daley CL, Grzemska M, Higashi JM, Ho CS, Hopewell PC, Keshavjee SA, Lienhardt C, Menzies R, Merrifield C, Narita M, O'Brien R, Peloquin CA, Raftery A, Saukkonen J, Schaaf HS, Sotgiu G, Starke JR, Migliori GB, Vernon A. Official American Thoracic Society/Centers for Disease Control and Prevention/Infectious Diseases Society of America Clinical Practice Guidelines: Treatment of Drug-Susceptible Tuberculosis. Clin Infect Dis. 2016 Oct 1;63(7):e147-e195. doi: 10.1093/cid/ciw376. Epub 2016 Aug 10. PMID 27516382
- [Background] Petrucci R, Lombardi G, Corsini I, Bacchi Reggiani ML, Visciotti F, Bernardi F, Landini MP, Cazzato S, Dal Monte P. Quantiferon-TB Gold In-Tube Improves Tuberculosis Diagnosis in Children. Pediatr Infect Dis J. 2017 Jan;36(1):44-49. doi: 10.1097/INF.0000000000001350. PMID 27749653
- [Background] Barcellini L, Borroni E, Brown J, Brunetti E, Codecasa L, Cugnata F, Dal Monte P, Di Serio C, Goletti D, Lombardi G, Lipman M, Rancoita PM, Tadolini M, Cirillo DM. First independent evaluation of QuantiFERON-TB Plus performance. Eur Respir J. 2016 May;47(5):1587-90. doi: 10.1183/13993003.02033-2015. Epub 2016 Feb 11. No abstract available. PMID 26869677
- [Background] Dorman SE, Schumacher SG, Alland D, Nabeta P, Armstrong DT, King B, Hall SL, Chakravorty S, Cirillo DM, Tukvadze N, Bablishvili N, Stevens W, Scott L, Rodrigues C, Kazi MI, Joloba M, Nakiyingi L, Nicol MP, Ghebrekristos Y, Anyango I, Murithi W, Dietze R, Lyrio Peres R, Skrahina A, Auchynka V, Chopra KK, Hanif M, Liu X, Yuan X, Boehme CC, Ellner JJ, Denkinger CM; study team. Xpert MTB/RIF Ultra for detection of Mycobacterium tuberculosis and rifampicin resistance: a prospective multicentre diagnostic accuracy study. Lancet Infect Dis. 2018 Jan;18(1):76-84. doi: 10.1016/S1473-3099(17)30691-6. Epub 2017 Nov 30. PMID 29198911
- [Background] Lombardi G, Di Gregori V, Girometti N, Tadolini M, Bisognin F, Dal Monte P. Diagnosis of smear-negative tuberculosis is greatly improved by Xpert MTB/RIF. PLoS One. 2017 Apr 21;12(4):e0176186. doi: 10.1371/journal.pone.0176186. eCollection 2017. PMID 28430807
- [Background] Internal Clinical Guidelines Team (UK). Tuberculosis: Prevention, Diagnosis, Management and Service Organisation. London: National Institute for Health and Care Excellence (UK); 2016 Jan. Available from http://www.ncbi.nlm.nih.gov/books/NBK338750/ PMID 26820019
- [Background] Jensen PA, Lambert LA, Iademarco MF, Ridzon R; CDC. Guidelines for preventing the transmission of Mycobacterium tuberculosis in health-care settings, 2005. MMWR Recomm Rep. 2005 Dec 30;54(RR-17):1-141. PMID 16382216
- [Background] Aliberti S, Codecasa LR, Gori A, Sotgiu G, Spotti M, Di Biagio A, Calcagno A, Nardini S, Assael BM, Tortoli E, Besozzi G, Ferrarese M, Matteelli A, Girardi E, De Lorenzo S, Seia M, Gramegna A, Del Prato B, Terranova L, Oriano M, Sverzellati N, Mirsaeidi M, Chalmers JD, Haworth CS, Loebinger MR, Aksamit T, Winthrop K, Ringshausen FC, Previdi G, Blasi F; IRENE Network. The Italian registry of pulmonary non-tuberculous mycobacteria - IRENE: the study protocol. Multidiscip Respir Med. 2018 Aug 9;13(Suppl 1):33. doi: 10.1186/s40248-018-0141-8. eCollection 2018. PMID 30151192
- [Background] Fattorini L, Mustazzolu A, Borroni E, Piccaro G, Giannoni F, Cirillo DM; Italian Multicentre Study on Resistance to Antituberculosis Drugs (SMIRA) Group. Tuberculosis in migrants from 106 countries to Italy, 2008-2014. Eur Respir J. 2016 Apr;47(4):1273-6. doi: 10.1183/13993003.01844-2015. Epub 2016 Feb 4. No abstract available. PMID 26846829
- [Background] Lombardi G, Dal Monte P, Denicolo A, Tadolini M, Martelli G, Bacchi Reggiani ML, Viale P, Landini MP. Trend of microbiologically-confirmed tuberculosis in a low-incidence setting with high immigration rates. BMC Public Health. 2014 Apr 10;14:340. doi: 10.1186/1471-2458-14-340. PMID 24721236
- See also: Agenzia Sanitaria e Sociale Regionale della Regione Emilia-Romagna. Epidemiologia della tubercolosi in Emilia-Romagna 2010-11. — https://assr.regione.emilia-romagna.it/pubblicazioni/rapporti-documenti/epidemiologia-della-tubercolosi-in-emilia-romagna-2010-2011-1
- See also: World Health Organization. Guidelines for the treatment of drug-susceptible tuberculosis and patient care (2017 update) — http://apps.who.int/iris/bitstream/10665/255052/1/9789241550000-eng.pdf?ua=1